CLINICAL TRIAL: NCT04198545
Title: Ethnic Differences in Iron Absorption
Brief Title: Ethnic Differences in Iron Absorption (FeGenes)
Acronym: FeGenes
Status: Active, not recruiting | Type: Observational
Sponsor: Cornell University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB # 1904008754; R01DK122216 (NIH)
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Anemia, Iron Deficiency; Iron Overload
Keywords: Iron absorption; Genetics
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Overload

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum and DNA samples will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to; 1) investigate population differences in iron absorption between East Asians and Northern Europeans; 2) assess population differences in hormonal and biochemical determinants of Fe absorption between East Asians and Northern Europeans; and 3) to investigate genetic contributions to Fe absorption, Fe status and Fe regulatory hormones between East Asians and Northern Europeans.

DETAILED DESCRIPTION:
Detailed description:

This study will utilize a multidisciplinary approach to identify genetic variation in genes that control iron utilization in order to shed light on the genetic basis of population differences in iron status and disease susceptibility with a long-term goal of informing population-specific dietary iron intake recommendations to minimize the risk of chronic diseases. To evaluate iron utilization, we will employ an in vivo, functional approach using an oral stable iron isotope method. Each participant will have genetic ancestry and genotyping evaluated using the Illumina Global Diversity Array-8. Study participants (n=504, aged 18-50 y) will consume 57Fe (as ferrous sulfate) in the fasted state and will then ingest a standardized breakfast and lunch meal. Two weeks after iron dosing, a blood sample will be collected from each participant and the amount of 57Fe incorporated into red blood cells will be measured using magnetic sector thermal ionization mass spectrometry. This project will fundamentally advance our understanding of ethnic differences in nutrient metabolism and iron status. It will also provide information to assist with the long-term goal of reducing the public health burden of Fe-related diseases.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Age between 18- 50y
* Non-smoking
* Not taking vitamin or mineral supplements.
* Females: premenopausal and not pregnant or lactating
* No preexisting medical complications (such as eating disorders, hemoglobinopathies, malabsorption diseases, steroid use, substance abuse history, or taking medications known to influence iron homeostasis)
* Body mass index (BMI) between 18 - 30 kg/m2.

Exclusion Criteria:

* BMI <18 or > 30 kg/m2,
* Age <18 y or > 50y,
* Not of Northern European or East Asian ancestry
* Smoking
* Pregnancy, lactating
* Have gastrointestinal disorders/malabsorption diseases/hemoglobinopathies/dietary restrictions/steroid use/ medication use of medications known to impact iron status, iron utilization or inflammatory status
* Take vitamin and mineral supplementations

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults from Ithaca and Rochester, NY
Sampling Method: Non-Probability Sample
Enrollment: 515 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The percent of non-heme iron absorption | 2-week
  The percent of non-heme iron absorption will be determined by red blood cell iron incorporation of stable 57Fe
The concentrations of iron and micronutrient status indicators | baseline and two-weeks post dosing
  The concentrations or serum folate, B12, hemoglobin, hematocrit, transferrin receptor, hepcidin, erythropoietin, erythroferrone, ferritin, interleukin-6, and c-reactive protein
Genetic ancestry and characterization of iron-related genotypes | baseline
  The DNA will be extracted from whole blood samples and each participant will have genetic ancestry and genotyping evaluated using the Illumina Global Diversity Array-8.
Habitual dietary information | baseline
  Habitual dietary information will be obtained from Diet History Questionnaire III .
Dietary information on the study day | baseline
  Detailed dietary information about all foods and beverages consumed on the study day will be obtained from the Automated Self-Administered 24-Hour Dietary Assessment Tool.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly O O'Brien, Principal Investigator — Cornell University
Locations (2):
- United States (2):
  - Cornell University, Ithaca, New York
  - University of Rochester, Rochester, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park CY, Barad A, Xu Y, Bender E, Thomas AK, Haller CM, Gu Z, Pressman EK, O'Brien KO. Dietary intake in East Asian and Northern European participants from the FeGenes study. Eur J Nutr. 2025 Jun 5;64(5):205. doi: 10.1007/s00394-025-03730-w. PMID 40471375
- [Derived] Barad A, Xu Y, Bender E, Pressman EK, Gu Z, O'Brien KO. Differences in nonheme iron absorption between healthy adults of East Asian or Northern European ancestry from the Iron Genes in East Asian and Northern European Adults Study (FeGenes): A cross-sectional stable iron isotope study. Am J Clin Nutr. 2025 Feb;121(2):417-426. doi: 10.1016/j.ajcnut.2024.11.015. PMID 39909711
- [Derived] Barad A, Xu Y, Bender E, Pressman EK, Gu Z, O'Brien KO. Iron regulatory hormones and their associations with iron status biomarkers among healthy adults of East Asian or Northern European ancestry: A cross-sectional comparison from the Iron Genes in East Asian and Northern European Adults Study (FeGenes). Am J Clin Nutr. 2025 Feb;121(2):406-416. doi: 10.1016/j.ajcnut.2024.10.018. PMID 39909710
- [Derived] Barad A, Xu Y, Bender E, Kang W, Xu R, Gu Z, Pressman EK, O'Brien KO. Characterization of iron status biomarkers and hematological indices among young adults of East Asian or Northern European ancestry: A cross-sectional analysis from the Iron Genes in East Asian and Northern European Adults Study (FeGenes). Am J Clin Nutr. 2025 Feb;121(2):394-405. doi: 10.1016/j.ajcnut.2024.10.014. PMID 39909709